CLINICAL TRIAL: NCT01633320
Title: Non-invasive Assessment of Immediate Postoperative Analgesia Using Analgesia/Nociception Index (ANI): A Prospective and Observational Study
Brief Title: Non-invasive Assessment of Immediate Postoperative Analgesia Using Analgesia/Nociception Index (ANI)
Status: Completed | Type: Observational
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Emmanuel Boselli, MD, PhD, Hôpital Edouard Herriot
Other Study IDs: CPP 2012-021 B
Record Dates: First submitted 2012-06-28; First posted 2012-07-04 (Estimated); Results first posted 2012-12-18 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-11

CONDITIONS: Postoperative Pain
Keywords: Analgesia/Nociception index
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to evaluate the clinical performance on Analgesia/Nociception Index (ANI) in the assessment of immediate postoperative analgesia in PACU in adult patients undergoing general anesthesia.

DETAILED DESCRIPTION:
Evaluation of the relationship between ANI and numerical rating pain scale (NRS) by linear regression.

Assessment of the performance of ANI to detect NRS>3 and NRS>=7 by building ROC curves.

ELIGIBILITY:
Inclusion Criteria:

* adult
* surgical or endoscopic procedures performed on general anesthesia

Exclusion Criteria:

* age <18 yrs or >75 yrs
* arrythmia
* administration of anticholinergic drugs or neuromuscular blockade reversal in the 20 previous minutes
* psychiatric diseases
* autonomic nervous system (ANS) disorders
* inability to understand the verbal rating pain scale.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients underoing surgical or endoscopic procedures performed on general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Bouvet, MD, Principal Investigator — Édouard Herriot hospital, HCL; Gérard Bégou, MD, Principal Investigator — Édouard Herriot hospital, HCL; Rabia Dabouz, MD, Principal Investigator — Édouard Herriot hospital, HCL; Christophe Magnin, MD, Principal Investigator — Édouard Herriot hospital, HCL; Bernard Allaouchiche, MD, PhD, Study Chair — Édouard Herriot hospital, HCL; Emmanuel Boselli, MD, PhD, Study Director — Édouard Herriot hospital, HCL; Mirela-Daniela Ionescu, MD, Principal Investigator — Édouard Herriot hospital, HCL
Locations (1):
- Department of Anesthesiology and Intensive Care, Édouard Herriot hospital, HCL, Lyon, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study performed between June and July 2012 at Édouard Herriot university hospital,Lyon, France.
  200 American Society of Anesthesiologists physical status I-II patients undergoing general anesthesia were included. The procedures performed were ear, nose and throat surgery or endoscopy and plastic surgery.
Pre-assignment Details: No patient were excluded from the trial before assignment to groups
Groups:
- NRS<=3 (no or Mild Pain): Patients with numerical rating pain scale <=3 at arrival in PACU
- NRS>3 (Moderate to Severe Pain): Patients with numerical rating scale pain score >3 at arrival in PACU
Period: Overall Study
Arm/Group | NRS<=3 (no or Mild Pain) | NRS>3 (Moderate to Severe Pain)
Started | 132 | 68
Completed | 132 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- NRS<=3: Patients with numerical rating scale <=3 at arrival in PACU
- NRS>3: Patients with numerical rating scale pain score >3 at arrival in PACU
- Total: Total of all reporting groups
Arm/Group | NRS<=3 | NRS>3 | Total
Number analyzed (Participants) | 132 | 68 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 118 | 62 | 180
  >=65 years | 14 | 6 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 41 (18) | 44 (15) | 43 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 26 | 88
  Male | 70 | 42 | 112
Region of Enrollment [Number; unit: participants]
  France | 132 | 68 | 200

OUTCOME MEASURES:

1. Primary Outcome: Analgesia/Nociception Index (ANI)
Description: The ANI is a 0-100 index estimating the parasympathetic/sympathetic balance derived from heart rate variability, measured by the PhysioDoloris monitor (MetroDoloris, Loos, France). High ANI values indicate parasympathetic predominance (no pain) while during nociception (increase in sympathetic activity), ANI value decrease to 60 or less.
Time Frame: At arrival in post-operative care unit (PACU) or 10 min after extubation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NRS<=3 | NRS>3
Number analyzed (Participants) | 132 | 68
units on a scale | 73 (17) | 49 (14)

2. Primary Outcome: Pain Scores on a 0-10 Numeric Rating Scale (NRS)
Description: Verbal pain scale, with 0 = no pain and 10 = worst pain imaginable. NRS<3 corresponds to no or mild pain NRS>=3 corresponds to moderate to severe pain NRS>=7 corresponds to severe pain
Time Frame: At arrival in PACU or 10 min after extubation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NRS<=3 | NRS>3
Number analyzed (Participants) | 132 | 68
units on a scale | 1 (1) | 5 (1)

ADVERSE EVENTS:
Arm/Group | NRS<=3 | NRS>3
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/68
Other Adverse Events (participants affected / at risk) | 0/132 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes